CLINICAL TRIAL: NCT06440538
Title: Improving Upper Limb Rehabilitation by Rebuilding Inter-limb Transfer of Motor Gains in Cervical SCI
Brief Title: Rebuilding Inter-limb Transfer in Cervical SCI
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: The Cleveland Clinic (Other)
Collaborators: The Craig H. Neilsen Foundation (Other)
Responsible Party: Principal Investigator, Ela B. Plow, Associate Proffesor, The Cleveland Clinic
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Supportive Care
Other Study IDs: 23-415
Record Dates: First submitted 2023-10-10; First posted 2024-06-04 (Actual); Last update posted 2025-09-24 (Actual); Status verified 2025-09

CONDITIONS: Cervical Spinal Cord Injury
Keywords: Cervical Spinal Cord Injury; Upper limb; Motor Training; Brain Stimulation; Peripheral Nerve Stimulation; Hand Dexterity; Inter-limb transfer; Motor learning

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (3):
- PCMS + Contralateral Motor Training (Experimental)
  Interventions: Device: PCMS + Contralateral Motor Training
- PCMS + Rest (Active Comparator)
  Interventions: Device: PCMS + Rest
- Sham PCMS + Contralateral Motor Training (Sham Comparator)
  Interventions: Device: Sham PCMS + Contralateral Motor Training

INTERVENTIONS:
Device: PCMS + Contralateral Motor Training — PCMS + Contralateral Motor Training will involve delivering 360 pairs of TMS-PNS pulses (30min, 0.2 Hz) to the weaker first dorsal interosseous (FDI) muscle immediately before a session of ballistic index finger abduction training at the opposite, stronger FDI muscle.
  Arms: PCMS + Contralateral Motor Training
Device: PCMS + Rest — PCMS + Rest will involve delivering 360 pairs of TMS-PNS pulses (30min, 0.2Hz) to the weaker FDI followed by a 30-min rest.
  Arms: PCMS + Rest
Device: Sham PCMS + Contralateral Motor Training — 360 TMS pulses will be delivered at a location 10-cm posterior to the participant's head (into the air, 0.2Hz) and no PNS pulses will be generated, followed by a session of 30-min ballistic index finger abduction training at the opposite, stronger FDI muscle.
  Arms: Sham PCMS + Contralateral Motor Training

SUMMARY:
The purpose of this study in people living with cervical Spinal Cord Injury (SCI) is to examine the effects of paired neurostimulation (i.e., PCMS) combined with contralateral motor training on inter-limb transfer of ballistic motor and hand dexterity skills.

DETAILED DESCRIPTION:
Cervical spinal cord injury (SCI) is the most common and severe type of SCI that can lead to paralysis of the trunk and all four limbs, also known as tetraplegia. People with tetraplegia place a high priority on regaining upper limb motor function to be independent in daily life. Despite intensive therapies, upper limb motor gains are slow to emerge, especially in chronic cases.

A critical barrier to effective and efficient upper limb rehabilitation in cervical SCI lies in the motor deficits of inter-limb transfer. Inter-limb transfer refers to a natural innate process within the human neuromotor system that motor skills acquired in one limb can transfer to the opposite, untrained limb, and is believed to play a key role in maximizing and accelerating post-injury recovery. Inter-limb transfer however is deficient following cervical SCI due to a breakdown of inter-limb neural connections at the cortical and spinal levels. Prior studies in uninjured people reveal that one can upregulate inter-limb neural mechanisms and hence augment inter-limb transfer effects by giving neurostimulation to augment corticomotoneuronal pathways to the untrained arm just before motor training in the contralateral arm.

This study aims to rebuild inter-limb transfer of motor gains in chronic cervical SCI using a novel non-invasive neurostimulation method called paired corticospinal-motor neuronal stimulation (PCMS). We will test the central hypothesis that PCMS given to an untrained hand immediately before the visuomotor ballistic motor training at the other hand will improve inter-limb transfer of ballistic motor and dexterity skills to the untrained hand, based on potentiation of inter-limb neural mechanisms.

ELIGIBILITY:
Inclusion Criteria:

* Neurological Level of Injury C4, C5, C6, C7, C8
* American Spinal Injury Association Impairment Scale (AIS) C-D
* greater than or equal to 1 year time post injury
* residual motor sparing of bilateral FDI muscles, defined as medical research council (MRC) grade 2 to 5

Exclusion Criteria:

* contraindications to transcranial magnetic stimulation (TMS) and peripheral nerve stimulation (PNS) including pacemaker, metal in the skull, seizure history, pregnancy, etc.
* history of alcohol and/or drug abuse
* current usage of medications that can potentially lower the seizure threshold such as bupropion, amphetamines, etc.
* history of other neurological conditions such as stroke, Parkinson's, and traumatic brain injury (TBI)
* active pressure ulcers to avoid disruption of ongoing medical treatments
* participation of on-going upper-limb therapies to minimize confounding effects
* excessive tone/spasticity (Modified Ashworth Scale [MAS] >3) and severe contractures or soft tissue shortening at elbow/wrist/fingers

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 17 (Estimated)
Dates: Start 2024-02-15 (Actual); Primary Completion 2026-07-30 (Estimated); Study Completion 2026-07-30 (Estimated)

PRIMARY OUTCOMES:
Change in ballistic acceleration | Baseline to post paired TMS and PNS stimulation, assessed for approximately 4-6 hours
  Participants perform 10 trials of ballistic index finger abduction with a accelerometer attached to index finger to capture the peak acceleration during the movement.
Change in excitability of cortical and corticospinal physiology and interhemispheric connections (TMS) | Baseline to post paired TMS and PNS stimulation, assessed for approximately 4-6 hours
  Transcranial magnetic stimulation will be used to test cortical output from both hemispheres and will be measured as motor evoked potentials(MEPS) of the First Dorsal Interosseous (FDI) muscle.
Change in excitability of spinal physiology (F-wave) | Baseline to post paired TMS and PNS stimulation, assessed for approximately 4-6 hours
  Peripheral Nerve stimulation will be performed to collect the spinal F-wave amplitude of the First Dorsal Interosseous (FDI) muscle.

SECONDARY OUTCOMES:
Change in Nine Hole Peg Test (NHPT) | Baseline to post paired TMS and PNS stimulation, assessed for approximately 4-6 hours
  The NHPT is used to measure finger dexterity measured in time to complete the test or amount of pegs placed in 100 sec.
Change in finger velocity smoothness during NHPT | Baseline to post paired TMS and PNS stimulation, assessed for approximately 4-6 hours
  The investigator will calculate the index finger(2nd digit) velocity smoothness using the number of local maxima of frontal plane finger velocities during the peg transfer phase using kinematic sensors place on the fingers.

OTHER OUTCOMES:
TMS safety questionnaire | Post paired TMS and PNS stimulation, assessed for approximately 4-6 hours
  A TMS safety questionnaire will be asked at the end of each TMS testing session
Capabilities of Upper Extremity Test(CUE-T) | Baseline
  CUE-T is a functional measure which identifies the functional ability of the upper limbs and is widely used in studies recruiting Spinal Cord Injury patients
Canadian Occupational Performance Measure (COPM) | Baseline
  COPM is used to measure participation restrictions of Spinal Cord Injury Subjects
Graded Redefined Assessment of Strength, Sensation and Prehension (GRASSP) | Baseline
  GRASSP is a functional measure which identifies the functional ability of the upper limbs and is widely used in studies recruiting Spinal Cord Injury patients
Spinal Cord Independence Measure(SCIM) | Baseline
  SCIM is a spinal cord injury measure that identifies activity limitations of self-care
Leisure Time Physical Activity Questionnaire for People with Spinal Cord Injury (LTPAQ-SCI) | Baseline
  The LTPAQ-SCI is an SCI-specific, self-report assessment of LTPA that measures the number of minutes of mild, moderate, and heavy exercises performed throughout a typical week.
Edinburgh Handedness Inventory | Baseline
  Questionnaire to ascertain the handedness of a participant in activities of daily living (ADL).

CONTACTS AND LOCATIONS:
Overall Officials: Ela Plow, PhD, Principal Investigator — The Cleveland Clinic
Locations (1):
- Lerner Research Institute; Cleveland Clinid Foundation, Cleveland, Ohio, United States